CLINICAL TRIAL: NCT00263445
Title: Constructing an Insulin-Like Growth Factor-based Prediction Model
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Pinchas Cohen, Proffessor and Chief, Peds Endo, University of California, Los Angeles
Other Study IDs: 04-07-052-02; 304-F02/X3270n (Genentech)
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Growth Hormone Deficiency; Idiopathic Short Stature; Small for Gestational Age
Keywords: Growth hormone dosing; IGF-I
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Serum insulin-like growth factor-I (IGF-I) measurements have been shown to correlate well with growth hormone action and effect, and recent data show that serum IGF-I may be related to safety and efficacy of growth hormone (GH) treatment in patients. Some studies indicate that high IGF-I levels are associated with increased cancer risk, and low IGF-I levels are associated with increased risk for cardiovascular disease. Studies in children also show that the serum IGF-I level is correlated with the change in height score achieved (that is, the higher the IGF-I level, the greater the gain in height). Pediatric endocrinologists have therefore begun to use serum IGF-I levels, in addition to growth rate and weight gain, to adjust the GH dose in treated children.

Although monitoring of serum IGF-I levels is becoming standard of care in patients begin treated with GH, there are few guidelines regarding the actual logistics of adjusting GH dose. As serum IGF-I level has been linked to both safety and efficacy of GH treatment, the ideal practice would be to maintain serum IGF-I levels within a certain target range. The overall goal of our study is to construct a mathematical model which predicts the change in GH dose necessary to achieve a desired change in IGF-I level.

Hypotheses to be tested by our study include the following: IGF-I measurement has a role in optimization of GH therapy; GH dose change to achieve IGF-I changes are predictable; and gender and puberty affect the relationship between dose change and target IGF-I changes.

DETAILED DESCRIPTION:
The first phase of our study, previously approved by the UCLA IRB in August 2004, involved a retrospective chart review and collection of preexisting data. We analyzed charts of patients who underwent non-weight-based GH dose adjustments preceded and followed by a serum IGF-I level. Data collected included patient's age, gender, height, weight, linear height velocity, pubertal status, GH dose, IGF-I levels, disease condition (i.e., growth hormone deficiency, idiopathic short stature, small-for-gestational age) and recording of any adverse effects. Based on this data collected, we performed statistical analysis of the relationship between GH dose change and change in IGF-I level achieved, and have found that in prepubertal children, there is a significant relationship between the GH dose change and change in corresponding IGF-I level. We have subsequently constructed a mathematical prediction model that allows us to determine the GH dose change necessary to achieve a desired IGF-I level, and in this second phase of our study, we plan to apply this mathematical prediction model prospectively for guiding GH dose adjustments in prepubertal children being treated with GH therapy.

Children being treated with GH are typically followed in the outpatient Endocrinology clinic every 3-4 months, and our practitioners have routinely been obtaining serum IGF-I levels (via venipuncture in the outpatient laboratory) for monitoring purposes. Validation of our GH dose change/IGF-I change prediction model will require assessment of sequential serum IGF-I level measurements immediately preceding a GH dose change, and again within 1-4 months following the GH dose change. We plan to continue our retrospective and ongoing analysis of patients who have paired values of GH dose adjustments preceded and followed by a serum IGF-I level, in order that we may continue to fine-tune our prediction model for optimizing GH dose adjustments.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal patients,
* Male/female,
* Ages 3-14 yrs,
* Being treated with growth hormone for the conditions of growth hormone deficiency, idiopathic short stature, and small-for-gestational age with failure to catch up to the normal growth curve by age 2 years.

Exclusion Criteria:

* Patients being treated with growth hormone for other conditions such as Turner syndrome, chronic renal failure, or Prader-Willi syndrome

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: GH-treated chlidren
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Delta IGF-I SDS | 3-months
  1 SDS change per 20% dose change

CONTACTS AND LOCATIONS:
Overall Officials: Pinchas Cohen, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Pediatric Endocrinology, Los Angeles, California, United States